CLINICAL TRIAL: NCT01967888
Title: A Phase 2/3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Assignment Study to Assess the Efficacy and Safety of Reparixin in Pancreatic Islet Auto-transplantation
Brief Title: Efficacy and Safety of Reparixin in Pancreatic Islet Auto-transplantation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REP0112
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Pancreatectomy for Chronic Pancreatitis
Keywords: Pancreatic islet auto-transplantation
MeSH Terms: interventions — reparixin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reparixin (Experimental): Solution for intravenous (IV) infusion with active compound
  Interventions: Drug: Reparixin
- Placebo (Placebo Comparator): Physiologic solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Reparixin — Solution for intravenous (IV) infusion; 2.772 mg/kg body weight/hour administered at 0.25 mL/kg/hour
  Other Names: DF1681Y
  Arms: Reparixin
Drug: Placebo — Physiologic solution administered at 0.25 mL/kg/hour
  Arms: Placebo

SUMMARY:
The study is a phase 2/3, multicenter, double-blind, parallel assignment study. It involves 100 adult recipients of an intra-hepatic pancreatic Islet Auto-Transplantation (IAT).

The objective of this clinical trial is to assess whether reparixin leads to improved transplant outcome as measured by the proportion of insulin-independent patients following IAT. The safety of reparixin in the specific clinical setting will be also evaluated.

DETAILED DESCRIPTION:
In contrast to allo-transplantation in type 1 diabetes patients, where immunological mechanisms involving allo- and auto-antibodies affect long-term graft function, outcome in IAT (Islet Auto-Transplantation) is independent from immunological processes and does not require immunosuppression management. On the other hand, early inflammatory events intrinsic to the intra-portal islet infusion have been demonstrated to impact islet engraftment. Among possible mechanisms, PMNs have been found to be the predominant cell types infiltrating the liver in a syngeneic model of islet transplantation in mice.

Data obtained in experimental models of islet transplantation in mice demonstrate a clear effect of reparixin in improving graft survival and function. Protection from the loss and/or deterioration of transplanted islets was evident regardless of the immunological mechanisms involved in islet damage, suggesting that the ability of reparixin to modulate early inflammatory responses readily impact graft outcome.

Thus, the use of reparixin may emerge as a potential useful medication in the control of non specific inflammatory events surrounding the early phases of IAT.

The goal of this study is to reach a total of 100 adult patients who are randomized and receive IAT after total or completion pancreatectomy. Patients will be randomly (1:1) assigned to receive either reparixin [continuous i.v. infusion for 7 days (168hrs)], or matched placebo (control group),starting approximately 12hrs before islet infusion. The two groups will be balanced within each centre. All patients who are randomized and receive the Investigational Product (either reparixin or placebo) will be included in the ITT analysis. Patients will be in the ITT analysis whether or not they receive IAT, because exclusions cannot be made for events occurring after randomization that could be influenced by the randomized assignment.

Recruitment will be competitive among the study sites, until the planned number of patients is enrolled. Competitive recruitment has been chosen to increase the speed of recruitment and to account for any difference in transplant rate among study sites. Each centre will enroll patients as rapidly as possible, up to a maximum of 40 patients (as per the randomization list). A maximum of 48 patients is allowed for the site of the Primary Investigator.

Each patient will be involved in the study for 7 day hospital stay during pancreatectomy followed by islet transplantation, for all required measurements up to hospital discharge and for 2 post-transplant visits scheduled @ day 75+14 and 365+14 after the transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for an IAT following total (or completion) pancreatectomy.
* Ages > 18 years.
* Patients willing and able to comply with the protocol procedures for the duration of the study, including scheduled follow-up visits and examinations.
* Patients who have given written informed consent, prior to any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.

Exclusion Criteria:

* Recipients of a previous IAT (if completion pancreatectomy).
* Patients undergoing total pancreatectomy due to either pancreatic cancer or pancreatic benign diseases other than chronic pancreatitis, including insulinomas, etc.
* Patients with inadequate renal reserve as per calculated creatinine clearance (CLcr) < 60 mL/min according to the Cockcroft-Gault formula (1976).
* Patients with hepatic dysfunction as defined by increased ALT/AST > 3 x upper limit of normal (ULN) or increased total bilirubin above the upper limit at local laboratory). Patients with Gilbert's syndrome (elevated unconjugated bilirubin levels in the absence of any evidence of hepatic or biliary tract disease) are not excluded.
* Patients with a preoperative International Normalized Ratio (INR) > 1.5 or any known coagulopathy.
* Hypersensitivity to:

  1. ibuprofen or to more than one non steroidal anti-inflammatory drug (NSAID).
  2. medications belonging to the class of sulfonamides, such as sulfamethazine, sulfamethoxazole, sulfasalazine, nimesulide or celecoxib.
* Concurrent sepsis (as per positive blood culture(s) and/or fever associated with other signs of systemic sepsis syndrome).
* Treatment with systemic steroids in the 2 weeks prior to enrolment (except for the use of <5mg prednisone daily or equivalent dose of hydrocortisone, for physiological replacement only) or with any immune modulators in the 4 weeks prior to enrolment.
* Patients with pre-existing diabetes or evidence of impaired β-cells function, based on pre-operative fasting blood glucose >115 mg/dL and/or a HbA1c > 6.5%, or requiring treatment with any anti-diabetic medication (e.g. insulin, metformin, etc) within the 2 weeks prior to enrolment.
* Use of any investigational agent in the 4 weeks prior to enrolment, including any anti-cytokine/chemokine agents.
* Pregnant or breast-feeding women; unwillingness to use effective contraceptive measures (females and males). (NB: pregnancy should be avoided in patients or partners during the first month after completing the treatment with the Investigational Product; no other specific warnings are described, considering the treatment course of the Investigational Product, its PK profile, and the lack of significant adverse effects on mating performance and fertility in animal studies).
* Patients with past or current history of alcohol abuse based on clinical history and/or past treatment for alcohol addiction.
* Patients with evidence of pre-operative portal hypertension as per clinical history and abdominal/liver imaging by ultrasound techniques.

Sites will comply with any additional or more restrictive exclusion criteria locally accepted, as per centre practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melena Bellin, MD, Principal Investigator — Schulze Diabetes Institute; University of Minnesota Amplatz Children's Hospital
Locations (9):
- United States (8):
  - University of California. Department of Surgery, Division of Transplantation, San Francisco, California
  - The University of Chicago Medical Center, Chicago, Illinois
  - Schulze Diabetes Institute University of Minnesota Medical School, Minneapolis, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - The University of Cincinnati Medical Center, Cincinnati, Ohio
  - Thomas E. Starzl Transplantation Institute University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas
- University of Alberta, Clinical Islet Transplant Program, Edmonton, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reparixin | Placebo
Started | 52 | 52
Completed | 42 | 45
Not Completed | 10 | 7
Not completed — Lost to Follow-up | 6 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Did Not Have Transplant | 1 | 0
Not completed — Research visit not done, data recorded | 1 | 0
Not completed — Subject excluded after randomization | 1 | 0
Not completed — Patient didn't proceed to pancreatectomy | 0 | 1
Not completed — Subject Unable To Comply With Final Day | 0 | 1

BASELINE CHARACTERISTICS:
Population: Two patients initially randomised to Reparixin received no treatment, hence were not included in the in the population analysed for demographics
Groups:
- Total: Total of all reporting groups
Arm/Group | Reparixin | Placebo | Total
Number analyzed (Participants) | 50 | 52 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 46 | 52 | 98
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (14.4) | 39.0 (10.0) | 39.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 38 | 71
  Male | 17 | 14 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 49 | 49 | 98
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 3 | 7
  United States | 46 | 49 | 95

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Were Insulin Independent After Islet Autotransplantation (IAT) at Day 365±14 Days After Transplant.
Description: Insulin-independence is defined as freedom from the need to take exogenous insulin for 14 or more consecutive days, with adequate glycemic control, as defined by:
  * a glycated hemoglobin (HbA1c) level <6.5%;
  * fingerstick fasting blood glucose not exceeding 126 mg/dL more than three times in the past week (based on a minimum of one daily measurement;
  * a 2 hour post-prandial blood glucose not exceeding 180 mg/dL more than four times in the past week (based on a minimum of one daily measurement);
  * a laboratory fasting glucose in the non-diabetic range (<126 mg/dL).
Time Frame: day 365±14 after the transplant
Population: ITT Population consists of all patients who were randomized and received the Investigational Product (either reparixin or placebo). Summarization and analysis of this population is based on randomized treatment, regardless of treatment actually received.
  Eligible patients are included in this population whether or not they receive IAT.
Measure: Number; unit: Percentage of participants
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 50 | 52
Percentage of participants | 20.0 | 21.2
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.542, Cochran-Mantel-Haenszel; t-test = -1.2, 95% CI 2-sided [-14.3 to 000]

2. Secondary Outcome: Area Under the Curve (AUC) for the Serum C-peptide Level at Day 75±14 After the Transplant
Description: AUC for the serum C-peptide level is calculated during the first 4 hours of an MMTT, normalized by the number of Islet Equivalent (IEQ)/kg
Time Frame: day 75±14 after the transplant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (ng/mL)/(IEQ/kg)*1000
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 43 | 48
(ng/mL)/(IEQ/kg)*1000 | 0.5314796 (0.3520819) | 0.6827533 (0.4769178)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.092, t-test, 2 sided; least square mean difference = -0.1601778, 95% CI 2-sided [-0.3178030 to -0.0025525]

3. Secondary Outcome: Area Under the Curve (AUC) for the Serum C-peptide Level at Day 365±14 After the Transplant
Description: AUC for the serum C-peptide level is calculated during the first 4 hours of a mixed meal tolerance test (MMTT), normalized by the number of Islet Equivalent (IEQ)/kg
Time Frame: day 365±14 after the transplant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (ng/mL)/(IEQ/kg)*1000
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 33 | 41
(ng/mL)/(IEQ/kg)*1000 | 0.5563432 (0.3133415) | 0.6865954 (0.4464460)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.161, t-test, 2 sided; least square mean difference = -0.1178242, 95% CI 2-sided [-0.2874310 to 0.0517825]

4. Secondary Outcome: Average Daily Insulin Requirements at Day 75±14 After the Transplant
Description: Daily insulin is reported as IU/kg and intake averaged over the previous week.
Time Frame: day 75±14 after the transplant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/kg/day
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 44 | 49
IU/kg/day | 0.2125 (0.1643) | 0.2190 (0.1589)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.846, t-test, 2 sided; least square mean difference = 0.0136, 95% CI 2-sided [-0.0508 to 0.0781]

5. Secondary Outcome: Average Daily Insulin Requirements at Day 365±14 After the Transplant
Description: Daily insulin is reported as IU/kg and intake averaged over the previous week.
Time Frame: day 365±14 after the transplant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/kg/day
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 39 | 43
IU/kg/day | 0.1723 (0.1893) | 0.1823 (0.1994)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.817, t-test, 2 sided; least square mean difference = -0.025, 95% CI 2-sided [-0.0939 to 0.0689]

6. Secondary Outcome: Time Course From Basal to 240 Min of Glucose Derived From the Mixed Meal Tolerance Test (MMTT) at Day 75±14 After the Transplant
Description: Data of this outcome are reported as "model estimates over all timepoints".
  This parameter was assessed at the following timepoints on the following numbers of patients for Reparixin and placebo, respectively:
  * basal; N=43; 48 (Basal is: 2 basal samples taken separately between -20 to 0 minutes before the meal followed by samples through 240 minutes after the meal).
  * 15 min; N=42; 46
  * 30 min; N=40; 46
  * 60 min; N=40; 46
  * 90 min; N=40; 46
  * 120 min; N=41; 46
  * 180 min; N=40; 46
  * 240 min; N=39; 44
Time Frame: day 75±14 after the transplant
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 50 | 52
mg/dL | 157.0894 (11.98160) | 166.5535 (11.45706)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.570, Mixed Models Analysis; least square mean difference = -9.4641, 95% CI 2-sided [-42.4900 to 23.5618]

7. Secondary Outcome: Time Course From Basal to 240 Min of Glucose Derived From the Mixed Meal Tolerance Test (MMTT) at Day 365±14 After the Transplant
Description: Data are reported as "model estimates over all timepoints"
  This parameters was assessed at the following timepoints on the following numbers of patients for Reparixin and placebo, respectively:
  * basal; N=34; 42 (Basal is: 2 basal samples taken separately between -20 to 0 minutes before the meal followed by samples through 240 minutes after the meal).
  * 15 min; N=34; 41
  * 30 min; N=34; 41
  * 60 min; N=34; 41
  * 90 min; N=34; 41
  * 120 min; N=34; 41
  * 180 min; N=33; 41
  * 240 min; N=33; 41
Time Frame: day 365±14 after the transplant
Population: ITT Population consists of all patients who were randomized and received the Investigational Product (either reparixin or placebo). Summarization and analysis of this population is based on randomized treatment, regardless of treatment actually received.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 50 | 52
mg/dL | 157.9988 (12.00455) | 180.9442 (12.08647)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.074, Mixed Models Analysis; least square mean difference = -22.9454, 95% CI 2-sided [-48.1826 to 2.2918]

8. Secondary Outcome: Time Course From Basal to 240 Min of C-peptide Derived From the Mixed Meal Tolerance Test (MMTT) at Day 75±14 After the Transplant
Description: Data are reported as "model estimates over all timepoints".
  This parameters was assessed at the following timepoints on the following numbers of patients for Reparixin and placebo, respectively:
  * basal; N=44; 48 (Basal is: 2 basal samples taken separately between -20 to 0 minutes before the meal followed by samples through 240 minutes after the meal).
  * 15 min; N=43; 47
  * 30 min; N=41; 47
  * 60 min; N=42; 47
  * 90 min; N=42; 47
  * 120 min; N=42; 47
  * 180 min; N=41; 47
  * 240 min; N=40; 44
Time Frame: day 75±14 after the transplant
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 50 | 52
ng/mL | 1.8976 (0.20787) | 2.1051 (0.20104)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.358, Mixed Models Analysis; least square mean difference = -0.2074, 95% CI 2-sided [-0.6538 to 0.2389]

9. Secondary Outcome: Time Course From Basal to 240 Min of C-peptide Derived From the Mixed Meal Tolerance Test (MMTT) at Day 365±14 After the Transplant
Description: Data are reported as "model estimates over all timepoints".
  This parameters was assessed at the following timepoints on the following numbers of patients for Reparixin and placebo, respectively:
  * basal; N=33; 41 (Basal is: 2 basal samples taken separately between -20 to 0 minutes before the meal followed by samples through 240 minutes after the meal).
  * 15 min; N=34; 41
  * 30 min; N=34; 41
  * 60 min; N=33; 41
  * 90 min; N=34; 41
  * 120 min; N=34; 41
  * 180 min; N=33; 40
  * 240 min; N=33; 41
Time Frame: day 365±14 after the transplant
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 50 | 52
ng/mL | 1.6052 (0.24507) | 1.8822 (0.24763)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.288, Mixed Models Analysis; least square mean difference = -0.2770, 95% CI 2-sided [-0.7936 to 0.2396]

10. Secondary Outcome: Time Course From Basal to 240 Min of Insulin Derived From the Mixed Meal Tolerance Test (MMTT) at Day 75±14 After the Transplant
Description: Data are reported as "model estimates over all timepoints".
  This parameter was assessed at the following timepoints on the following numbers of patients for Reparixin and placebo, respectively:
  * basal; N=43; 48 (Basal is: 2 basal samples taken separately between -20 to 0 minutes before the meal followed by samples through 240 minutes after the meal).
  * 15 min; N=43; 47
  * 30 min; N=41; 47
  * 60 min; N=41; 47
  * 90 min; N=41; 47
  * 120 min; N=42; 47
  * 180 min; N=41; 47
  * 240 min; N=40; 44
Time Frame: day 75±14 after the transplant
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: UIU/mL
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 50 | 52
UIU/mL | 23.67209 (3.497499) | 23.57493 (3.378854)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.980, Mixed Models Analysis; least square mean difference = 0.09716, 95% CI 2-sided [-7.41834 to 7.61266]

11. Secondary Outcome: Time Course From Basal to 240 Min of Insulin Derived From the Mixed Meal Tolerance Test (MMTT) at Day 365±14 After the Transplant
Description: Data are reported as "model estimates over all timepoints".
  This parameter was assessed at the following timepoints on the following numbers of patients for Reparixin and placebo, respectively:
  * basal; N=34; 41 (Basal is: 2 basal samples taken separately between -20 to 0 minutes before the meal followed by samples through 240 minutes after the meal)
  * 15 min; N=34; 41
  * 30 min; N=34; 41
  * 60 min; N=34; 41
  * 90 min; N=34; 41
  * 120 min; N=34; 41
  * 180 min; N=33; 41
  * 240 min; N=33; 40
Time Frame: day 365±14 after the transplant
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: UIU/mL
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 50 | 52
UIU/mL | 22.85522 (3.718512) | 21.77905 (3.757573)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.785, Mixed Models Analysis; least square mean difference = 1.07617, 95% CI 2-sided [-6.76562 to 8.91796]

12. Secondary Outcome: β-cell Function at Day 75±14 After the Transplant
Description: This variable is assessed by β-score (assessment of β-cell function after islet transplantation). The total score is calculated on a 0-8 scoring system (higher is a better outcome) that gives 0-2 points each for:
  * fasting plasma glucose,
  * HbA1c,
  * stimulated C-peptide
  * insulin requirement subscales. The higher the total score, the better the outcome.
  * Fasting (or before breakfast) plasma glucose (mg/dL) : ≤99, Score 2; 100-124, Score 1; ≥ 125, Score 0 (the higher the subscore the better the outcome)
  * HbA1c (%): ≤6.1, Score 2; 6.2-6.9, Score 1; ≥ 7.0, Score 0 (the higher the subscore the better the outcome)
  * Daily average (previous week) insulin (IU/kg/day): ---, Score 2; 0.01-0.24, Score 1; ≥ 0.25, Score 0 (the higher the subscore the better the outcome)
  * Stimulated C-peptide (ng/mL): ≥ 0.9, Score 2; 0.3-0.89, Score 1; ≤0.3, Score 0 (the higher the subscore the better the outcome)
Time Frame: day 75±14 after the transplant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 42 | 47
score on a scale | 5.7 (1.6) | 5.2 (1.9)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.176, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: β-cell Function at Day 365±14 After the Transplant
Description: This variable is assessed by β-score (assessment of β-cell function after islet transplantation). The total score is calculated on a 0-8 scoring system (higher is a better outcome) that gives 0-2 points each for glucose, HbA1c, stimulated C-peptide and insulin requirement subscales.
  The higher the total score the better the outcome.
  * Fasting (or before breakfast) plasma glucose (mg/dL) : ≤99, Score 2; 100-124, Score 1; ≥ 125, Score 0 (the higher the subscore the better the outcome)
  * HbA1c (%): ≤6.1, Score 2; 6.2-6.9, Score 1; ≥ 7.0, Score 0 (the higher the subscore the better the outcome)
  * Daily average (previous week) insulin (IU/kg/day): ---, Score 2; 0.01-0.24, Score 1; ≥ 0.25, Score 0 (the higher the subscore the better the outcome)
  * Stimulated C-peptide (ng/mL): ≥ 0.9, Score 2; 0.3-0.89, Score 1; ≤0.3, Score 0 (the higher the subscore the better the outcome)
Time Frame: day 365±14 after the transplant
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 32 | 41
score on a scale | 5.9 (2.0) | 5.4 (2.4)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.403, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Proportion of Patients With an HbA1c <6.5% at Day 365±14 After the Transplant
Description: Percentage of patients with a glycated haemoglobin (HbA1c) <6.5% at day 365±14 after the transplant.
Time Frame: day 365±14 after the transplant
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 42 | 45
percentage of participants | 64.3 [49.79 to 78.78] | 62.2 [48.06 to 76.39]
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.842, Chi-squared; Treatment effect = 2.1, 95% CI 2-sided [-18.20 to 22.33]

15. Secondary Outcome: Cumulative Number of Severe Hypoglycemic Events From Day 75±14 to Day 365±14 After the Transplant
Description: A severe hypoglycemic event is defined as an event with one of the following symptoms: "memory loss, confusion, uncontrollable behavior, irrational behavior, unusual difficulty in awakening, suspected seizure, seizure, loss of consciousness, or visual symptoms", in which the subject was unable to treat him/herself and which was associated with either a blood glucose level <54mg/dL or prompt recovery after oral carbohydrate, i.v. glucose, or glucagon administration.
Time Frame: from day 75±14 to day 365±14 after the transplant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 41 | 44
number of events | 0.1 (0.94) | 0.0 (0.21)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.339, Anderson-Gill model; Hazard Ratio (HR) = 3.21, 95% CI 2-sided [0.29 to 34.97]

16. Secondary Outcome: Proportion of Patients With an HbA1c <6.5% at Day 365±14 After the Transplant AND Free of Severe Hypoglycemic Events From Day 75±14 to Day 365±14 After the Transplant Inclusive
Description: Percentage of patients with an HbA1c <6.5% at day 365±14 after the transplant AND free of severe hypoglycemic events from day 75±14 to day 365±14 after the transplant inclusive.A severe hypoglycemic event is defined as an event with one of the following symptoms: "memory loss, confusion, uncontrollable behavior, irrational behavior, unusual difficulty in awakening, suspected seizure, seizure, loss of consciousness, or visual symptoms", in which the subject was unable to treat him/herself and which was associated with either a blood glucose level <54mg/dL or prompt recovery after oral carbohydrate, i.v. glucose, or glucagon administration.
Time Frame: from day 75±14 to day 365±14 after the transplant
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 39 | 44
percentage of participants | 64.1 [49.05 to 79.16] | 59.1 [44.56 to 73.62]
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.640, Chi-squared; Treatment effect = 5.0, 95% CI 2-sided [-15.91 to 25.93]

17. Secondary Outcome: Incidence and Severity of Adverse Events and Serious Adverse Events Throughout the Study
Description: The percentages of patients with any treatment emergent adverse events (TEAE, serious and non serious) and with serious TEAE by severity are presented.
  Patients with multiple events within a particular system organ class or preferred term were counted only under the category of their most severe event within that system organ class or preferred term.
  A serious AE was defined as any untoward medical occurrence that at any dose:
  * Resulted in death
  * Was life-threatening (ie, the patient was at risk of death at the time of the event)
  * Required inpatient hospitalization or prolongation of existing hospitalization
  * Resulted in persistent or significant disability/incapacity
  * Was a congenital anomaly/birth defect
  * Was an important medical event that, based upon appropriate medical judgment, may have jeopardized the patient and may have required medical or surgical intervention to prevent one of the outcomes listed above
Time Frame: up to day 365±14 after the transplant
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 50 | 52
percentage of patients
  TEAE- Mild events | 90.0 | 92.3
  TEAE - Moderate events | 90.0 | 80.8
  TEAE - Severe events | 64.0 | 53.8
  serious TEAE- Mild events | 18.0 | 23.1
  serious TEAE- Moderate events | 22.0 | 13.5
  serious TEAE- Severe events | 42.0 | 32.7

18. Secondary Outcome: Proportion of Patients Falling Into One of the Following Malnutrition Risk Levels (Poor Prognosis, Significant Risk, Increased Risk, Normal) According to Pre-albumin Level at Day 75±14 After the Transplant
Description: Malnutrition risk levels are defined as:
  * Poor prognosis = pre-albumin level <5.0 mg/dL
  * Significant risk = pre-albumin level 5.0 to 10.9 mg/dL
  * Increased risk = pre-albumin level 11.0 to 15.0 mg/dL
  * Normal = pre-albumin level > 15.0 (up to 35.0) mg/dL
Time Frame: day 75±14 after the transplant
Population: Safety Population consists of all randomized patients. Summarization and analysis of this population was based on treatment actually received. Patients randomized but not treated were analyzed in the total summary statistics only.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 42 | 46
percentage of patients
  poor prognosis | 0 [0.00 to 8.41] | 0 [0.00 to 7.71]
  significant risk | 9.5 [2.66 to 22.62] | 4.3 [0.53 to 14.84]
  increased risk | 45.2 [29.85 to 61.33] | 28.3 [15.99 to 43.46]
  normal | 45.2 [29.85 to 61.33] | 67.4 [51.98 to 80.47]

19. Secondary Outcome: Proportion of Patients Falling Into One of the Following Malnutrition Risk Levels (Poor Prognosis, Significant Risk, Increased Risk, Normal) According to Pre-albumin Level at Day 365±14 After the Transplant
Description: as for outcome 18
Time Frame: day 365±14 after the transplant
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 40 | 44
percentage of participants
  Poor prognosis | 5.0 [0.61 to 16.92] | 0 [0.00 to 8.04]
  Significant risk | 2.5 [0.06 to 13.16] | 6.8 [1.43 to 18.66]
  Increased risk | 27.5 [14.60 to 43.89] | 9.1 [2.53 to 21.67]
  Normal | 65.0 [48.32 to 79.37] | 84.1 [69.93 to 93.36]

20. Secondary Outcome: Proportion of Patients by Steatorrhea Severity at Day 75±14 After the Transplant
Description: Levels of steatorrhea severity (evaluated in the 4 weeks prior to day 75±14 and 365±14), are defined as:
  * No steatorrhea;
  * Steatorrhea few times per week;
  * Steatorrhea daily;
  * Stool incontinence.
Time Frame: day 75±14 after the transplant
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 44 | 48
percentage of participants
  no steatorrhea | 54.5 [38.85 to 69.61] | 64.6 [49.46 to 77.84]
  steatorrhea few times per week | 29.5 [16.76 to 45.20] | 25.0 [13.64 to 39.60]
  steatorrhea daily | 11.4 [3.79 to 24.56] | 6.3 [1.31 to 17.20]
  stool incontinence | 4.5 [0.56 to 15.47] | 4.2 [0.51 to 14.25]

21. Secondary Outcome: Proportion of Patients by Steatorrhea Severity at Day 365±14 After the Transplant
Description: as for outcome 20
Time Frame: day 365±14 after the transplant
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 42 | 46
percentage of participants
  no steatorrhea | 52.4 [36.42 to 68.00] | 58.7 [43.23 to 73.00]
  steatorrhea few times per week | 26.2 [13.86 to 42.04] | 19.6 [9.36 to 33.91]
  steatorrhea daily | 21.4 [10.30 to 36.81] | 21.7 [10.95 to 36.36]
  stool incontinence | 0 [0.00 to 8.41] | 0 [0.00 to 7.71]

22. Secondary Outcome: Cumulative Number of Episodes of Documented Asymptomatic Hypoglycemia From Day 75±14 to Day 365±14 After the Transplant
Description: The following definition applies:
  - Asymptomatic hypoglycemia = An event not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose concentration <70mg/dL.
Time Frame: from day 75±14 to day 365±14 after the transplant
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 41 | 45
number of episodes | 1.5 (4.3) | 4.4 (25.6)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.448, Wilcoxon rank-sum test

23. Secondary Outcome: Cumulative Number of Episodes of Documented Symptomatic Hypoglycemia From Day 75±14 to Day 365±14 After the Transplant
Description: The following definition applies:
  - Documented symptomatic hypoglycemia = An event during which typical symptoms of hypoglycemia are accompanied by a measured plasma glucose concentration <70mg/dL.
Time Frame: from day 75±14 to day 365±14 after the transplant
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 41 | 45
number of episodes | 4.6 (13.9) | 4.8 (17.8)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.910, Wilcoxon rank-sum test

24. Secondary Outcome: Cumulative Number of Diabetic Ketoacidosis-related Events
Description: A diabetic ketoacidosis event is defined as the presence of:
  * hyperglycemia (blood glucose >200 mg/dL);
  * pH <7.3 or HCO3 <15;
  * ketones positive in the serum or urine.
Time Frame: from day 75±14 to day 365±14 after the transplant
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 41 | 46
number of events | 0.0 (0.0) | 0.0 (0.0)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 1.000, Wilcoxon rank-sum test

25. Secondary Outcome: Peak C-peptide at Day 75 After the Transplant
Description: Peak C-peptide (C-P) is a known predictor of Type 1 Diabetes.
Time Frame: Day 75±14 after the transplant
Population: ITT population: ITT Population consists of all patients who were randomized and received the Investigational Product (either reparixin or placebo). Summarization and analysis of this population is based on randomized treatment, regardless of treatment actually received.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 44 | 48
ng/mL | 2.640 (1.529) | 2.900 (1.753)

26. Secondary Outcome: Peak C-peptide at Day 365 After the Transplant
Description: Peak C-peptide (C-P) is a known predictor of Type 1 Diabetes.
Time Frame: Day 365±14 after the transplant
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 34 | 41
ng/mL | 2.630 (1.467) | 3.170 (1.843)

27. Secondary Outcome: Time-to-peak C-peptide at Day 75 After the Transplant
Description: The time-to-peak value in minutes was computed as the time of the peak value (HH:MM on a 24-hour clock) minus the end time of the mixed meal (HH:MM on a 24-hour clock) as recorded on the mixed meal tolerance test Case Report Form.
Time Frame: day 75±14 and day 365±14 after the transplant
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 43 | 44
minutes | 104.2 (93.6) | 108.7 (59.4)

28. Secondary Outcome: Time-to-peak C-peptide at Day 365 After the Transplant
Description: The time to peak value in minutes will be computed as the time of the peak value (HH:MM on a 24-hour clock) minus the end time of the mixed meal (HH:MM on a 24-hour clock) as recorded on the mixed meal tolerance test CRF.
Time Frame: Day 365±14 after the transplant
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 31 | 40
minutes | 97.8 (90.9) | 102.0 (56.2)

29. Secondary Outcome: Change From Baseline in Post-transplant Alanine Aminotransferase (ALT)
Description: Data are reported as "model estimates over all timepoints".
  This safety parameter was assessed at the following timepoints on the following numbers of patients for Reparixin and placebo, respectively:
  * baseline; N=50; 52
  * Day 2 post-transplant; N=49; 51
  * Day 3 post-transplant; N=47; 50
  * Day 7 post-transplant; N=47; 50
  * Day 75 post-transplant; N=44; 47
Time Frame: Baseline, Days 2, 3, 7, 75 ±14 after the transplant
Population: Safety Population: Safety Population consists of all randomized patients. Summarization and analysis of this population was based on treatment actually received. Patients randomized but not treated.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 50 | 52
U/L | 60.4105 (40.9699) | 29.0615 (40.2724)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.5018, Mixed Models Analysis; least square mean difference = 31.3491, 95% CI 2-sided [-60.9980 to 123.70]

30. Secondary Outcome: Change From Baseline in Post-transplant Aspartate Aminotransferase (AST)
Description: as for outcome 29
Time Frame: Baseline, Days 2, 3, 7, 75±14 after the transplant
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 50 | 52
U/L | 46.8755 (27.8248) | 23.3301 (26.6545)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.4537, Mixed Models Analysis; Least square mean difference = 23.5454, 95% CI 2-sided [-38.6619 to 85.7528]

31. Secondary Outcome: Number of Treatment Emergent Adverse Events Related to Investigational Product
Description: Treatment emergent adverse events - possibly, probably and highly probably - related to investigational product are called "Adverse reactions" (ADR).
  An adverse reaction is defined as any untoward medical occurrence in a patient or clinical investigation patient, which has a causal relationship with the administered medicinal product.
Time Frame: Throughout the study From Day -1 to hospital discharge
Population: Safety Population:Safety Population consists of all randomized patients. Summarization and analysis of this population was based on treatment actually received. Patients randomized but not treated were analyzed in the total summary statistics only.
Measure: Number; unit: Number of events
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 50 | 52
Number of events
  possibly related | 20 | 28
  probably related | 0 | 0
  highly probably related | 0 | 0

32. Secondary Outcome: Number of Serious Treatment Emergent Adverse Events Related to Investigational Product
Description: Serious Treatment emergent adverse events - possibly, probably and highly probably - related to investigational product are called serious "Adverse reactions".
  A serious adverse reaction is defined as any untoward medical occurrence with a causal relationship with the administered medicinal product, that at any dose:
  * Resulted in death
  * Was life-threatening (ie, the patient was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it were more severe.)
  * Required patient hospitalization or prolongation of existing hospitalization
  * Resulted in persistent or significant disability/incapacity
  * Was an important medical event that, based upon appropriate medical judgment, may have jeopardized the patient and may have required medical or surgical intervention to prevent one of the outcomes listed above
Time Frame: Throughout the study From Day -1 to hospital discharge for all adverse events, and from then to day 365 post-transplantation only for serious adverse events
Population: Safety population: Safety Population consists of all randomized patients. Summarization and analysis of this population were based on treatment received. Patients randomized but not treated were analyzed in the total summary statistics only.
Measure: Number; unit: Number of events
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 50 | 52
Number of events
  possibly related | 4 | 1
  probably related | 0 | 0
  highly probably related | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day -1 to hospital discharge for all adverse events, and from then to day 365 post-transplantation only for serious adverse events.
Arm/Group | Reparixin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/52
Serious Adverse Events (participants affected / at risk) | 29/50 | 30/52
Other Adverse Events (participants affected / at risk) | 46/50 | 48/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reparixin (N=50) | Placebo (N=52)
Abdominal pain (Gastrointestinal disorders) | 13 (22) | 7 (19)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (7)
Nausea (Gastrointestinal disorders) | 3 (4) | 4 (10)
small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (8)
abdominal hernia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Haemorrage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrintestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
impaired gastric empting (Gastrointestinal disorders) | 1 (1) | 0 (0)
intestinal ischeamia (Gastrointestinal disorders) | 0 (0) | 1 (1)
omental infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Urinary tract infections (Infections and infestations) | 2 (2) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 2 (3) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Gastrenteritis viral (Infections and infestations) | 0 (0) | 1 (2)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Joint abscess (Infections and infestations) | 0 (0) | 1 (1)
postoperative abscess (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroparesis postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post operative hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (6) | 2 (4)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 1 (2)
Hernia (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Vascular stent occlusion (General disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Depressed levele of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Migrane (Nervous system disorders) | 0 (0) | 1 (2)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 2 (3) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Leucocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Mental status changes (Psychiatric disorders) | 1 (2) | 0 (0)
Confusion of state (Psychiatric disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reparixin (N=50) | Placebo (N=52)
Procedural pain (Injury, poisoning and procedural complications) | 37 (37) | 43 (43)
Incision site pain (Injury, poisoning and procedural complications) | 5 (7) | 2 (3)
Procedural nausea (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 22 (23) | 19 (22)
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 (11) | 14 (14)
Hypoglycaemia (Metabolism and nutrition disorders) | 10 (12) | 11 (12)
Hypophosphataemia (Metabolism and nutrition disorders) | 9 (9) | 12 (12)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 (7) | 6 (6)
Hypernatraemia (Metabolism and nutrition disorders) | 6 (6) | 4 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hypoinsulinaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypervolaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Vitamin C deficiency (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Calcium deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin A deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 19 (26) | 21 (21)
Abdominal pain (Gastrointestinal disorders) | 8 (10) | 3 (3)
Constipation (Gastrointestinal disorders) | 11 (11) | 16 (16)
Vomiting (Gastrointestinal disorders) | 8 (8) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 3 (3)
Ileus (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bile acid malabsorption (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jejunal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
mesenteric artery trhombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 25 (25) | 22 (22)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorragic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (5)
Penumonia (Infections and infestations) | 0 (0) | 4 (4)
Clostridium difficile infection (Infections and infestations) | 3 (3) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 3 (3)
Abdominal infection (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1)
Respiratory moniliasis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 1 (1)
Haematocrit decreased (Investigations) | 2 (2) | 2 (2)
Haemoglobin decreased (Investigations) | 2 (2) | 2 (2)
Oxygen saturation decreased (Investigations) | 1 (1) | 3 (3)
Urin output decreased (Investigations) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Bacterial test positive (Investigations) | 0 (0) | 3 (3)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
Blood potassium decreased (Investigations) | 2 (2) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 3 (3)
White blood cell count increased (Investigations) | 0 (0) | 3 (3)
Mean arterial pressure decreased (Investigations) | 1 (1) | 1 (1)
Protein total decreased (Investigations) | 1 (1) | 1 (1)
Blood creatinin decreased (Investigations) | 0 (0) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1)
Blood alkalyne phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0)
Blood zinc decreased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Catheter culture positive (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Fibrin degradation products increased (Investigations) | 0 (0) | 1 (1)
International normalized ratio increased (Investigations) | 1 (1) | 0 (0)
Portal vein pressure increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 10 (13) | 10 (11)
Oedema peripheral (General disorders) | 1 (1) | 3 (3)
Pain (General disorders) | 2 (3) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (3)
Asthenia (General disorders) | 0 (0) | 1 (1)
Breackthrough pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Generalized oedema (General disorders) | 1 (1) | 0 (0)
Secretion discharge (General disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 10 (10) | 12 (13)
Hypertension (Vascular disorders) | 7 (9) | 4 (4)
Anxiety (Psychiatric disorders) | 4 (4) | 11 (11)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7) | 6 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rush (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Thachycardia (Cardiac disorders) | 4 (4) | 9 (9)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disk degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular wickness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ìHeadache (Nervous system disorders) | 0 (0) | 3 (3)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Stupor (Nervous system disorders) | 1 (1) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Dyisuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Non reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT01967888/Prot_003.pdf
  • Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT01967888/SAP_000.pdf